CLINICAL TRIAL: NCT01114191
Title: Ph I Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Linifanib (ABT-869)
Brief Title: A Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Linifanib (ABT-869)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Mark McKee, MD, Medical Director, Oncology, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M11-306
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — linifanib; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: ABT-869; Drug: ketoconazole

INTERVENTIONS:
Drug: ABT-869 — 2.5mg [5 mg days 1, 8 and 12. 17.5 mg on days 13 and after]
  Other Names: linifanib, ABT-869
Drug: ketoconazole — 400 mg days 6-11

SUMMARY:
This is a phase 1, open-label study designed to determine the interaction of ketoconazole with ABT-869.

DETAILED DESCRIPTION:
This study is designed to explore the drug interaction between ketoconazole and ABT-869 to determine the potential effect of ketoconazole on the metabolism of ABT-869. ABT-869 will be taken alone or in combination with ketoconazole. The safety of a single dose administration of ABT-869 when administered alone and in combination with ketoconazole will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Male or female and age is >= 18 years.
2. Must have a histologically or cytologically confirmed non-hematologic malignancy.
3. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
4. Must have adequate bone marrow, renal and hepatic function as follows:

   * Bone Marrow: Absolute neutrophil count (ANC) >= 1,500/mm3; Platelets >= 100,000/mm3 ; Hemoglobin >= 9.0 g/dL
   * Renal function: serum creatinine <= 2.0 mg/dL;
   * Hepatic function: AST and ALT <= 1.5 x ULN unless liver metastases are present, then AST and ALT <= 5.0 x ULN; bilirubin <= 1.5 mg/dL
5. Must have PTT <= 1.5 x ULN and/or INR <= 1.5.
6. Women of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 90 days following completion of therapy. Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

   * Total abstinence from sexual intercourse (minimum one complete menstrual cycle);
   * Vasectomized male subjects or vasectomized partner of female subjects;
   * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration; if the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after study completion;
   * Intrauterine device (IUD);
   * Double barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or creams);
   * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completion of therapy.
7. Is capable of understanding and complying with parameters as outlined in the protocol and able to sign the informed consent, approved by an Independent Ethic Committee (IEC)/Institutional Review Board (IRB) prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria

1. Has received anti-cancer therapy including investigational agents, cytotoxic chemotherapy, radiation therapy or biologic therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to study drug administration. In addition subject has not recovered to less than or equal to Grade 1 clinically significant adverse effects/toxicities of the previous therapy.
2. Has undergone major surgery within 21 days of Study Day 1.
3. Has untreated brain or meningeal metastases. Subjects with treated brain metastases that are radiographically or clinically stable (for at least 4 weeks after therapy) and who have no evidence of cavitation or hemorrhage in the brain lesion, are eligible provided that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to Study Day 1).
4. Has a central thoracic tumor lesion as defined by location involving or abutting the hilar structures. The presence of central nodal disease is allowed.
5. Female subjects who are pregnant or breastfeeding.
6. Has received potential inhibitors of the metabolism of linifanib within 21 days prior to initial study drug administration. Such drugs include CYP3A inhibitors e.g., triazole, itraconazole, ketoconazole, fluconazole, grapefruit juice, verapamil, diltiazem, aprepitant, clarithromycin and erythromycin; CYP1A2 inhibitors e.g., fluvoxamine, ciprofloxacin, mexiletine, propafenone and zileuton; CYP2C19 inhibitors e.g., omeprazole; CYP2C8 substrates e.g., repaglinide, paclitaxel and rosiglitazone and CYP3A inducers e.g., rifampin and carbamazepine.
7. Has proteinuria defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade > 1 at baseline as measured by a urine dipstick (2+ or greater) and confirmed by a 24 hour urine collection (> 1 g/24 hrs). Subjects may be re-screened if proteinuria is shown to be controlled with or without intervention.
8. Currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (BP) > 100 mmHg; or systolic blood pressure (BP) > 150 mmHg. Subjects may be re-screened if BP is shown to be controlled with or without intervention.
9. Clinically significant uncontrolled condition(s) including but not limited to:

   * Active uncontrolled infection
   * Class III or IV heart failure as defined by the New York Heart Association functional classification system
   * Unstable angina pectoris or cardiac arrhythmia
   * Myocardial infarction within last 6 months
   * History of adrenal insufficiency
   * History of cerebral vascular accident within last 6 months
   * Active ulcerative colitis, Crohn's disease, celiac disease or any other conditions that interfere with absorption
   * History of autoimmune disease with kidney involvement
   * History of overt bleeding (> 30 mL bleeding/episode) within 3 months of study drug administration
   * Psychiatric illness/social situation that would limit compliance with study requirements
   * Any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities
10. Is receiving combination anti-retroviral therapy for human immunodeficiency virus (HIV).
11. Has consumed grapefruit or grapefruit products within 21 days prior to initial study drug administration.
12. Has a documented left ventricular (LV) ejection fraction < 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of ketoconazole on the pharmacokinetics of ABT-869 in subjects with advanced or metastatic solid tumors. | Different timepoints on Days 1-12
  Blood samples for the PK of ABT-869 and ketoconazole will be collected at designated time points throughout the study.

SECONDARY OUTCOMES:
Safety: Adverse Events - The number of participants with adverse events will be reported as a measure of Safety. | Throughout the study
  Adverse event monitoring, lab tests assessments, physical exam and vital signs will be evaluated throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D McKee, MD, Study Director — Abbott
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 35784, Detroit, Michigan
  - Site Reference ID/Investigator# 36527, Lebanon, New Hampshire